CLINICAL TRIAL: NCT06231953
Title: A Prospective, Multi-center Clinical Study to Establish Multi-Cancer Early Detection Platform Through the Analysis of Whole Genome Sequencing of Circulating DNA in Cancer Patients and Healthy Volunteers.
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0299
Record Dates: First submitted 2023-05-18; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Invasive Cancer; Healthy Volunteer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients: Patients who have diagnosed as invasive cancers
- Healthy volunteers: Subjects who have done cancer screening tests

SUMMARY:
This is a prospective, multi-center clinical study of Multi-Cancer Early Detection (MCED) testing in cancer patients and healthy volunteers. The purpose of this study is to establish MCED platform through the analysis of whole genome sequencing of circulating DNA.

The study will enroll 4,000 subjects as defined by eligibility criteria at up to 10 clinical institutions in South Korea.

DETAILED DESCRIPTION:
AIMA is analysing whole genome sequencing data of circulating tumor DNA, combined through machine learning technique, to develop MCED platform to detect early stage cancer.

The purpose of this prospective, multi-center, observational study is to validate an MCED platform for the early detection of cancers.

The investigators will collect blood samples from subjects who are diagnosed as invasive cancers before treatment or from healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years or older
* Subjects who have been diagnosed with stages 1 to 4 of solid tumor or healthy volunteers who have scheduled a cancer screening examination
* Subjects who have agreed to provide clinical information and blood samples
* Subjects who have agreed for the storage and secondary use of residual blood samples for research
* Subjects who have understood the study and are able to provide a written informed consent

Exclusion Criteria:

* Subjects who are not appropriate for the study because of intellectual disabilities or severe mental disorders
* Subjects with a history of HIV, HTLV, or Syphilis infection
* Subjects with primary site unknown cancer or synchronous or metachronous double primary cancers
* Subjects who have diagnosed with any other malignant tumor within the past 5 years (except for cured non-melanoma skin cancer, in situ cancer, or thyroid cancer)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have diagnosed invasive cancer or healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of invasive cancer, assessed by positive predictive value and negative predictive value | 36 months
Accuracy of prediction for the origin of cancer, assessed by concordance rate | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Joohyuk Sohn, Principal Investigator — Division of Medical Oncology, Yonsei Cancer Center, Yonsei Univ. College of Medicine
Locations (1):
- Yonsei Cancer Center, Yonsei Univ. College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No